CLINICAL TRIAL: NCT01924507
Title: Intensive Cared Bedside Sleep Medicine
Brief Title: Bedside Sleep Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Fatima Dumas Cintra, MD, PhD, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bedsidesleep; AFIP (Other Grant/Funding Number: AFIP)
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Sleep Disorders; Sleep Apnea; Acute Myocardial Infarction; Acute Decompensated Heart Failure
Keywords: Sleep medicine; Sleep apnea; Acute myocardial infarction; Heart failure; CPAP
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): Patients with apnea will be treated with CPAP during the night.
  Interventions: Device: CPAP
- Control (No Intervention): One arm group will be control and will not receive CPAP treatment during the ICU admission.

INTERVENTIONS:
Device: CPAP — CPAP - continuous positive air pressure in patients with sleep apnea
  Arms: CPAP

SUMMARY:
The investigators aimed to evaluated the role of bedside sleep medicine in an cardiology intensive care unit. The patients will be submitted to a overnight polysomnography. Those individuals with sleep apnea will be treated with CPAP during the ICU admission. Also, the investigators will identify the factors that compromise the sleep and will act to minimize them to improve the sleep quality.

After the interventions, the investigators will evaluate if there are reduced days of hospital admission, major cardiovascular events (infarction, reinfarction, heart failure and stroke) and overall mortality.

DETAILED DESCRIPTION:
At the hospital discharge and after at 1, 3 and 12 months we will evaluate the occurrence of major cardiovascular events (infarction, reinfarction, heart failure and stroke) and overall mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Acute decompensated heart failure
* Age > 18 years-old
* Cardiology intensive care unit admission

Exclusion Criteria:

* Intravenous sedation
* Invasive mechanical ventilation
* hemodynamic instability
* use of intravenous vasoactive drugs
* acute respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
days of admission | 7 days
  Days of admission in the cardiology intensive care unit

SECONDARY OUTCOMES:
Combination of acute myocardial infarction, reinfarction, heart failure and stroke | 12 months

OTHER OUTCOMES:
Overall mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Paulo - Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Freedman NS, Kotzer N, Schwab RJ. Patient perception of sleep quality and etiology of sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1155-62. doi: 10.1164/ajrccm.159.4.9806141. PMID 10194160
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Aaron JN, Carlisle CC, Carskadon MA, Meyer TJ, Hill NS, Millman RP. Environmental noise as a cause of sleep disruption in an intermediate respiratory care unit. Sleep. 1996 Nov;19(9):707-10. doi: 10.1093/sleep/19.9.707. PMID 9122557
- [Background] Gami AS, Olson EJ, Shen WK, Wright RS, Ballman KV, Hodge DO, Herges RM, Howard DE, Somers VK. Obstructive sleep apnea and the risk of sudden cardiac death: a longitudinal study of 10,701 adults. J Am Coll Cardiol. 2013 Aug 13;62(7):610-6. doi: 10.1016/j.jacc.2013.04.080. Epub 2013 Jun 13. PMID 23770166
- [Background] Martinez-Garcia MA, Campos-Rodriguez F, Catalan-Serra P, Soler-Cataluna JJ, Almeida-Gonzalez C, De la Cruz Moron I, Duran-Cantolla J, Montserrat JM. Cardiovascular mortality in obstructive sleep apnea in the elderly: role of long-term continuous positive airway pressure treatment: a prospective observational study. Am J Respir Crit Care Med. 2012 Nov 1;186(9):909-16. doi: 10.1164/rccm.201203-0448OC. Epub 2012 Sep 13. PMID 22983957
- [Background] Elliott R, McKinley S, Cistulli P. The quality and duration of sleep in the intensive care setting: an integrative review. Int J Nurs Stud. 2011 Mar;48(3):384-400. doi: 10.1016/j.ijnurstu.2010.11.006. Epub 2010 Dec 24. PMID 21185560
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100